CLINICAL TRIAL: NCT06655844
Title: Extended Home-use Trial of a Novel Device to Reduce Chronic Pain
Brief Title: Sana Device for Post-Treatment Lyme Disease Syndrome Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Sana Health, Inc. (Unknown)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-18-01103
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Post-treatment Lyme Disease Syndrome; Chronic Pain
MeSH Terms: conditions — Post-Lyme Disease Syndrome; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Arm (Experimental): This group will experience the active device settings.
  Interventions: Device: Sana Pain Reliever
- Sham Arm (Sham Comparator): This group will experience the sham device settings.
  Interventions: Device: Sham SPR

INTERVENTIONS:
Device: Sana Pain Reliever — The Sana Pain Reliever (Sana PR) by Sana Health Inc is a device comprised of one (1) main component (Mask with Earbuds) and two (2) ancillary components (Charger and Headband). The device is worn over the eyes (with earbuds in ears).
  Arms: Real Arm
Device: Sham SPR — Participants will receive the SPR device and a tablet with instructions of how to use the device and how to answer the questionnaires on the tablet mobile application. Each session with the device will last 15 minutes and run under the device's sham settings. The session consists of periods of light and sounds (beeps). Participants will be instructed to use the device each day at the end of the day prior to going to sleep and whenever they experience heightened pain during the day.
  Arms: Sham Arm

SUMMARY:
This study will investigate the effectiveness of the Sana Pain Reliever (Sana PR) at reducing chronic pain.

The Sana PR is a device comprised of one main component (Mask with Earbuds) and two ancillary components (Charger and Headband). The device is worn over the eyes (with earbuds in ears). The device pulses light at a single wavelength but various frequencies throughout a specific firmware algorithm. Through the earbuds, the device also plays different tones in conjunction with the pulses. The device has a skin contacting Heart Rate Variability (HRV) sensor built into the forehead area that measures HRV throughout the use of the device.

The system runs for 15 min at a time and is not FDA approved.

The trial will last a total of 14 weeks.

50 participants who have a diagnosis of Post-treatment Lyme Disease and experience chronic pain are expected to take part in this study at Mount Sinai.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical diagnosis of neuropathic pain AND
* Confirmed clinical diagnosis of Post-treatment Lyme disease syndrome
* Diagnosis will be based on participants meeting either Group 1 or Group 2 criteria of the Columbia Clinical Trial Network PTLDS diagnostic criteria:

  * Group 1. Well-defined Lyme disease meeting CDC Surveillance Definition
  * Erythema Migrans
  * History of possible exposure to a high incidence county or state (or an adjacent area)
* Erythema migrans rash

  * EM 1: EM rash diagnosed by HCP previously (either in person or telemedicine)
  * EM 1A: MOA self-report & medical record documentation of rash > 5 cm
  * EM 1B: MOA: self-report and medical record documentation of EM rash but not size
  * EM 1C: MOA: self-report & rash misdiagnosed in medical record as cellulitis/spider bite
  * EM 1D: MOA: self-report and either: photo of EM or Class 1 lab test confirmation within 4 weeks of illness onset OR Disseminated "objective" manifestation with lab test confirmation of Bb infection
* Clinical history includes at least one of the following symptoms/signs, which are not better accounted for by another cause (MOA: medical records and/or self-report).
* Neurologic: Lymphocytic Meningitis; Encephalitis; Encephalomyelitis, Cranial Neuritis (especially facial palsy); Radiculoneuropathy;
* Other Neurologic Signs (with objective measures): Encephalopathy, Polyneuropathy
* Carditis: 2nd or 3rd degree AV block; Myocarditis; Pericarditis
* Lyme arthritis: Recurrent joint swelling in one or more joints
* Dermatologic: Disseminated EM ("satellite") or Acrodermatitis atrophicans AND
* Lab test Confirmation (previous) (requires at least one of the Class 1 lab tests) (MOA: self-report & documentation) Group 2. Probable.
* Chronic Multisystem Symptoms attributed to Lyme disease (insufficient to meet Group 1) and not better explained by another diagnosis and patient has evidence of positive lab results on a Class 1 lab test (or 4 of 10 bands for IgG Western blot (WB)) (MOA: self-report with lab documentation
* Class 1 lab test confirmation (excluding IgM WB)
* Highly suggestive IgG WB (4 of 10 bands) OR EM rash by history after exposure to a Lyme-endemic area but not previously diagnosed by a HCP and no photo or Class 1 lab test confirmation is available (MOA: self-report) OR Viral like illness (not better explained by other cause) with indeterminate or + enzyme immunoassay (EIA) with positive IgM WB or positive Class 1 lab test (within 4 weeks of illness onset after known exposure to a Lyme high-incidence area for standard two-tiered (STT) IgM) (MOA: medical records, lab test and self-report) (MOA: lab test and self-report) OR
* Viral like illness (not better explained by other cause) with indeterminate or positive EIA with positive IgM WB or positive Class 1 lab test (within 6 months of illness onset after known exposure to a Lyme high-incidence area for standard twotiered (STT) IgM) (MOA: medical records, lab test and self-report) (MOA: lab test and self-report)
* Ages 18+
* Fluent in English
* Consistent medications for the last 4 weeks prior to the first baseline visit (week 0)

Exclusion Criteria:

* Diagnosis of photosensitive epilepsy
* Ear or eye infection
* Vision impairments that affect perception of light in one or both eyes
* Deafness in one or both ears
* Psychiatric disorders (participants will not be excluded if they score 0-30 points on the BDI, or if participants self- report having anxiety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Symptom Inventory | Baseline 1 (Week 0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
  This scale was developed to assess both the quantitative and qualitative qualities of neuropathic pain (NP). It includes 12 items, assessing spontaneous pain, brief attacks of pain, provoked pain and abnormal sensations in the painful area. This is a sensitive tool for measuring changes in neuropathic pain after a therapeutic intervention. Full scale from 0-10 with higher score indicating more symptom. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline 1 (Week 0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. Full score from 0-21, with higher score indicating worse sleep quality. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Beck Depression Inventory (BDI) | Baseline 1 (Week 0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
  The Beck Depression Inventory (BDI) is used to evaluate depression symptoms, which are estimated to be highly prevalent in chronic pain populations. This questionnaire is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Depression may be a major contributor to a lack of reduction of pain. Scoring is from 0 (minimal) to 3 (severe), with total score from 0-63. Higher total scores indicate more severe depressive symptoms. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
General Anxiety Disorder 7-item questionnaire (GAD-7) | Baseline 1 (Week 0); Baseline 2 (Week 2); Post-assessment (Week 10); Follow up (Week 14)
  The General Anxiety Disorder 7-item questionnaire (GAD-7) is a 7-item questionnaire that asks user to rank how often they have been bothered by seven problems over the past two weeks from "0" (not at all) to "3" (nearly every day). The items that users are asked to rank levels of nervousness, anxiousness, relaxing, restlessness, irritability and fearfulness. Full scale from 0-21, with higher score indicating more symptoms. Change in score at Week 2, Week 10 and Week 14 as compared to Baseline.
Patient's Global Impression of Change (PGIC) | Post-assessment (Week 10); Follow up (Week 14)
  The Patient's Global Impression of Change (PGIC) will be used to assess self-reported relieving effect. It will evaluate pain from no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7). The patients will answer the following question: "Since beginning treatment at this program, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life related to your condition?". Full score from 0-7, with higher score indicating more improvement. Change in score at Week 14 as compared to Week 10.
Visual analogue scale (VAS)- Pain | VAS-Pain: before and after each time they use the device up to 14 weeks
  Visual Analog Scale (VAS) to measure pain: a measure of "no pain" to "Worst pain imaginable" along a line. Participants will be asked to mark the level of their pain along the line. Full scale from 0-100 with higher score indicating more pain.
Visual analogue scale (VAS)- Sleep | VAS-Sleep: once/day up to 14 Weeks
  Visual Analog Scale (VAS) to measure sleep: a measure of "did not sleep at all" to "best possible night's sleep" along a line. Participants will be asked to mark the level of their sleep along the line. The Sana Health application will prompt users to answer this scale before they use the device for the first time each day. Full scale from 0-10 with higher score indicating more pain.

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Cohen Center for Recovery from Complex Chronic Illnesses (CoRE), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD. Not applicable.